CLINICAL TRIAL: NCT00141440
Title: The Effect of Cycling Off Criteria During Pressure Support Ventilation in Chronic Obstructive Pulmonary Disease (COPD) Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Policlinico Hospital (Other)
Responsible Party: Davide Chiumello, Policlinico Hospital
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1073
Record Dates: First submitted 2005-08-31; First posted 2005-09-01 (Estimated); Last update posted 2009-12-30 (Estimated); Status verified 2008-09

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: gas exchange; pressure support ventilation; respiratory mechanics; COPD patients
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Respiration, Artificial

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): COPD patients
  Interventions: Procedure: mechanical ventilation

INTERVENTIONS:
Procedure: mechanical ventilation — evaluated the effect of two different cycling off criteria on breathing pattern, respiratory effort, and gas exchange in patients with chronic obstructive pulmonary disease

SUMMARY:
The investigators' aim is to study the effect of cycling off criteria during pressure support ventilation in COPD patients at two levels of PEEP and PSV.

DETAILED DESCRIPTION:
In this study two levels of cycling off criteria at two levels of PEEP and PSV were tested in term of gas exchange, respiratory mechanics, work of breathing and patient comfort.

ELIGIBILITY:
Inclusion Criteria:

* Stable COPD patients during invasive mechanical ventilation

Exclusion Criteria:

* Hemodynamic instability,
* Paralysis

Ages: 16 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2005-07; Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Respiratory mechanics, gas exchange | 2 minutes

SECONDARY OUTCOMES:
Comfort of breathing | 2 minutes

CONTACTS AND LOCATIONS:
Overall Officials: davide chiumello, md, Principal Investigator — Policlinico Hospital; Davide Chiumello, MD, Study Chair — Policlinico
Locations (1):
- Ospedale Sacco, Milan, milano, Italy

REFERENCES:
- [Result] Chiumello D, Polli F, Tallarini F, Chierichetti M, Motta G, Azzari S, Colombo R, Rech R, Pelosi P, Raimondi F, Gattinoni L. Effect of different cycling-off criteria and positive end-expiratory pressure during pressure support ventilation in patients with chronic obstructive pulmonary disease. Crit Care Med. 2007 Nov;35(11):2547-52. doi: 10.1097/01.CCM.0000287594.80110.34. PMID 17893630